CLINICAL TRIAL: NCT00313014
Title: A Multicenter, Randomized, Double-blind, Active Comparator Study to Determine the Efficacy and Safety of BTDS 20 or Oxycodone Immediate-release Versus BTDS 5 in Subjects With Moderate to Severe Low Back Pain
Brief Title: Safety and Efficacy of Buprenorphine Transdermal System (BTDS) in Subjects With Moderate to Severe Low Back Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated early due to administrative reasons unrelated to efficacy or safety.
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BUP3015
Record Dates: First submitted 2006-04-10; First posted 2006-04-11 (Estimated); Results first posted 2010-09-29 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Low back pain; opioid; transdermal; Butrans
MeSH Terms: conditions — Low Back Pain | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BTDS 5 (Active Comparator): Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear.
  Interventions: Drug: Buprenorphine
- BTDS 20 (Experimental): Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear.
  Interventions: Drug: Buprenorphine
- Oxycodone Immediate-Release (Experimental): Oxycodone immediate-release 40 mg (two 5-mg capsules every 6 hours).
  Interventions: Drug: Oxycodone Immediate-Release

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear.
  Other Names: Butrans™
  Arms: BTDS 5
Drug: Buprenorphine — Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear
  Other Names: Butrans™
  Arms: BTDS 20
Drug: Oxycodone Immediate-Release — Oxycodone HCl immediate-release 40 mg (two 5-mg capsules every 6 hours).
  Arms: Oxycodone Immediate-Release

SUMMARY:
The objective of this study is to demonstrate the effectiveness and tolerability of the buprenorphine transdermal system (BTDS) 20 in comparison to the buprenorphine transdermal system (BTDS) 5 and oxycodone immediate-release in subjects with moderate to severe low back pain currently treated with oral opioids. The double-blind treatment intervention duration is 12 weeks during which time supplemental analgesic medication (acetaminophen, ibuprofen) will be provided to all subjects in addition to study drug.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* low back pain for 3 months or longer, confirmed by radiographic evidence.
* receiving a stable dose of an opioid analgesic for low back pain.

Exclusion Criteria:

* taking more than 80 mg per day of oral morphine sulfate or equivalent within 30 days of enrollment.
* requiring frequent analgesic therapy for chronic condition(s), in addition to low back pain.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2004-02; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hale, MD, Principal Investigator — Gold Coast Research LLC, Weston, FL, USA
Locations (85):
- United States (85):
  - Birmingham Pain Center, Birmingham, Alabama
  - Arthritis Clinical Intervention Program, Birmingham, Alabama
  - Winston Physician Services, LLC, Haleyville, Alabama
  - Arizona Research Center, Inc., Phoenix, Arizona
  - Radiant Research, Phoenix, Arizona
  - Advanced Clinical Therapeutics, Tuscon, Arizona
  - Hot Springs Pain Clinic, Hot Springs, Arkansas
  - NuLife Clinical Research, Inc., Anaheim, California
  - Lovelace Scientific Resources, Inc., Beverly Hills, California
  - Northern California Research Corp, Carmichael, California
  - International Clinical Research Network, Chula Vista, California
  - Shreenath Clinical Service, Fountain Valley, California
  - U of Calif at Davis, Med Ctr, Pain Management Center, Sacramento, California
  - Accelovance, San Diego, California
  - Southern Colorado Clinic, Pueblo, Colorado
  - Chiefland Medical Center, Chiefland, Florida
  - University Clinical Research, Inc., DeLand, Florida
  - Drug Study Institute, Jupiter, Florida
  - Innovative Research of West Florida, Inc., Largo, Florida
  - Renstar Medical, Ocala, Florida
  - Peninsula Research Inc., Ormond Beach, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Coastal Medical Research, Port Orange, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Georgia Medical Research Institute, Marietta, Georgia
  - Atlanta Knee & Shoulder Clinic, Stockbridge, Georgia
  - Pain Care Boise, Boise, Idaho
  - Idaho Arthritis and Osteoporosis Center, Meridian, Idaho
  - Pain and Rehabilitation Clinic of Chicago, Chicago, Illinois
  - GFI Research Center, Evansville, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Medical Associates Clinics, Dubuque, Iowa
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - CTT, Inc., Prairie Village, Kansas
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - New Orleans Clinical Trial Management Inc., Metairie, Louisiana
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - Research Center of Louisiana, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Future Care Studies, Springfield, Massachusetts
  - Rheumatology PC, Kalamazoo, Michigan
  - Lake Michigan Clinical Research & Consulting, Inc., Saint Joseph, Michigan
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - HealthCare Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Lovelace Scientific Resources, Henderson, Nevada
  - Pivotal Research Centers, North Las Vegas, Nevada
  - Research Across America, New York, New York
  - Pain and Orthopedic Neurology , Charlotte Spine Center,, Charlotte, North Carolina
  - Metrolina Medical Research, Charlotte, North Carolina
  - Triangle Orthopaedic Associates, Durham, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - MedArk Clinical Research, Morgantown, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Odyssey Research, Bismarck, North Dakota
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Associated Medical Services, Oklahoma City, Oklahoma
  - Keystone Clinical Research, Altoona, Pennsylvania
  - Valley Pain Specialists, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Central Pennsylvania Clinical Research, Mechanicsburg, Pennsylvania
  - BioMedical Research Associates, Shippensburg, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - New England Center Clinical Research, Cranston, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Arthritis & Osteoporosis Center, Orangeburg, South Carolina
  - Brown Clinic, Watertown, South Dakota
  - Holston Medical Group, Bristol, Tennessee
  - Tri Cities Medical Research, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Galenos Research, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - Team Research of Central Texas, Harker Heights, Texas
  - KRK Medical Research, Richardson, Texas
  - Benchmark Research, San Angelo, Texas
  - Unlimited Research, San Antonio, Texas
  - Texas Medical Research Associates, San Antonio, Texas
  - Clinical Trial Network Oaks Medical Center, Spring, Texas
  - N. Texas Neuro Research, Wichita Falls, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Dean Medical Center, Oregon, Wisconsin

REFERENCES:
- [Result] Steiner D, Munera C, Hale M, Ripa S, Landau C. Efficacy and safety of buprenorphine transdermal system (BTDS) for chronic moderate to severe low back pain: a randomized, double-blind study. J Pain. 2011 Nov;12(11):1163-73. doi: 10.1016/j.jpain.2011.06.003. Epub 2011 Jul 31. PMID 21807566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began with first patient first visit (FPFV) on 25-Feb-2004 to last patient last visit (LPLV) on 23-Sep-2005, at 75 medical/research sites in the United States.
Pre-assignment Details: Prerandomization: screening period [Prospective assessment: subjects were assessed to ensure compliance with all inclusion/exclusion criteria]. Opioid taper segment: assessed the severity of the subject's low back pain upon analgesic medication discontinuation. Open-label run-in period: identified subjects whose pain was controlled with BTDS 20.
Groups:
- Double-blind BTDS 5: Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear
- Double-blind BTDS 20: Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear
- Double-blind Oxycodone Immediate-Release: Oxycodone HCl immediate-release 40 mg (two 5-mg capsules every 6 hours).
Period: Overall Study
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Started | 221 | 219 | 220
Completed | 128 | 146 | 159
Not Completed | 93 | 73 | 61
Not completed — Withdrawal by Subject | 11 | 7 | 5
Not completed — Adverse Event | 14 | 29 | 16
Not completed — Lost to Follow-up | 7 | 6 | 10
Not completed — Administrative | 9 | 6 | 14
Not completed — Lack of Efficacy | 52 | 25 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release | Total
Number analyzed (Participants) | 221 | 219 | 220 | 660
Age Continuous [Mean (Standard Deviation); unit: years] | 50.2 (12.88) | 50.4 (11.93) | 49.5 (12.37) | 50.0 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 113 | 100 | 314
  Male | 120 | 106 | 120 | 346

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Over the Last 24 Hours Score at Weeks 4, 8, and 12.
Description: Subjects were evaluated during the double-blind phase for "average pain over the last 24 hours" prior to the study visits. Pain scale is 11 points (0 = no pain to 10 = pain as bad as you can imagine)
Time Frame: Last 24 hours score at weeks 4, 8, 12 of the double-blind phase
Population: Full Analysis Population (N = 660) consisted of subjects who were randomized and received at least 1 dose of double-blind study drug.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Number analyzed (Participants) | 221 | 219 | 220
units on a scale
  Screening | 6.36 (0.075) | 6.46 (0.084) | 6.46 (0.079)
  Prerandomization | 2.84 (0.075) | 2.91 (0.075) | 2.74 (0.074)
  Week 4 | 3.79 (0.149) | 3.40 (0.128) | 3.14 (0.125)
  Week 8 | 3.83 (0.162) | 3.35 (0.140) | 3.24 (0.145)
  Week 12 | 4.02 (0.179) | 3.35 (0.139) | 3.26 (0.152)
Statistical Analysis 1: Comparison: Double-blind BTDS 5 vs Double-blind BTDS 20; The null hypothesis was that there was no difference between BTDS 20 or oxycodone HCl immediate-release 40 mg with respect to BTDS 5. The alternative hypothesis was that the BTDS 20 arm was different from the BTDS 5 arm; Test type: Superiority or Other; p < .001, Mixed Models Analysis — P value was 2-sided and performed at the 5% error level; Repeated measures mixed linear model with treatment, time, and time by treatment interaction as fixed effects; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-0.99 to -0.35], Standard Error of Mean 0.163
Statistical Analysis 2: Comparison: Double-blind BTDS 5 vs Double-blind Oxycodone Immediate-Release; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — P value was 2-sided and performed at the 5% error level; Repeated measures mixed linear model with treatment, time, and time by treatment interaction as fixed effect; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.07 to -0.44], Standard Error of Mean 0.161

2. Secondary Outcome: Mean Daily Number of Supplemental Analgesic Tablets
Description: The mean daily number of tablets of supplemental analgesic medications used during the double-blind phase
Time Frame: Double-blind phase (84 days)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: tablets
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Number analyzed (Participants) | 221 | 219 | 220
tablets | 3.8 (0.12) | 3.3 (0.13) | 3.5 (.13)
Statistical Analysis 1: Comparison: Double-blind BTDS 5 vs Double-blind BTDS 20; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .006, ANCOVA — To address the issue of multiplicity and control the family-wise error rate, a gate-keeping strategy and a stepwise approach (Holm's methodology) were used to evaluate the statistical significance of the secondary efficacy analyses; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.90 to -0.13] — The analysis was based on the number of subjects who took > 1 tablet of supplemental analgesia
Statistical Analysis 2: Comparison: Double-blind BTDS 5 vs Double-blind Oxycodone Immediate-Release; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .158, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.70 to 0.09] — The analysis was based on the number of subjects who took > 1 tablet of supplemental analgesia

3. Secondary Outcome: Oswestry Disability Index (ODI) Score (V 2.0)
Description: The ODI (version 2) is a low back pain-specific, validated instrument that consists of questions related to limitations in performing specific activities of daily living and 1 question related to pain intensity. The ODI is a self-administered questionnaire that is usually completed in less than 5 minutes.
  The ODI consists of 10 sections. Each section consists of 6 statements ranked from 0 to 5 (0 = good to 5 = worse). (Note: A higher score represents greater disability.)
Time Frame: Weeks 4, 8, 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Number analyzed (Participants) | 221 | 219 | 220
units on a scale
  Week 4 | 34.80 (1.066) | 33.04 (1.019) | 30.79 (1.124)
  Week 8 | 35.69 (1.245) | 34.27 (1.094) | 31.64 (1.165)
  Week 12 | 36.30 (1.392) | 33.06 (1.231) | 32.96 (1.243)
Statistical Analysis 1: Comparison: Double-blind BTDS 5 vs Double-blind BTDS 20; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .065, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-3.55 to 0.11]
Statistical Analysis 2: Comparison: Double-blind BTDS 5 vs Double-blind Oxycodone Immediate-Release; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .031, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.99, 95% CI [-3.79 to -0.18]

4. Secondary Outcome: The Sleep Disturbance Subscale in the MOS-Sleep Scale at Weeks 4, 8, and 12.
Description: The MOS-Sleep Scale consists of 12 individual items: (4 sleep disturbance, 2 sleep adequacy, 1 quantity/ optimal sleep, 3 somnolence, 1 snoring, and 1 shortness of breath).
  Question 1 is scored on a scale of 1 to 5 and Questions 3 to 12 are scored on a scale of 1 to 6. The Sleep Disturbance Subscale score is derived from the scores to Questions 1, 3, 7 and 8, and ranges from 0 to 100, where higher scores indicate greater sleep disturbance.
Time Frame: Weeks 4, 8, 12 of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release
Number analyzed (Participants) | 221 | 219 | 220
units on a scale
  Week 4 | 40.67 (2.025) | 34.65 (1.607) | 38.10 (1.788)
  Week 8 | 42.28 (2.264) | 35.69 (1.721) | 39.17 (1.924)
  Week 12 | 40.85 (2.376) | 33.65 (1.941) | 41.60 (2.205)
Statistical Analysis 1: Comparison: Double-blind BTDS 5 vs Double-blind BTDS 20; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mixed linear model: treatment, time as fixed effects, screening, prerandomization sleep disturbance subscale as covariates; subject as a random effect; Mean Difference (Final Values) = -6.23, 95% CI 2-sided [-9.64 to -2.82], Standard Error of Mean 1.735
Statistical Analysis 2: Comparison: Double-blind BTDS 5 vs Double-blind Oxycodone Immediate-Release; The null hypothesis was that there was no difference between BTDS 20 or oxycodone HCl immediate-release 40 mg with respect to BTDS 5. The alternative hypothesis was that BTDS 20 arm was different from the BTDS 5 arm; Test type: Superiority or Other; p = .121, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.65, 95% CI [-6.01 to 0.70], Standard Error of Mean 1.709

ADVERSE EVENTS:
Time Frame: Adverse events occurring after the signing of the informed consent up to end of study and 7 days after, discontinuation, or serious AEs occurring up to 30 days following the last study visit were followed until the AE or sequelae resolved or stabilized.
Description: AEs were learned of by spontaneous reports, subject interview, and daily diary.
Groups:
- Double-blind Oxycodone Immediate-Release: Oxycodone immediate-release 40 mg (two 5-mg capsules every 6 hours).
- Open-label Run-in Period, BTDS 10/20: Open-label BTDS 10 or 20 mcg/h applied for 7-day wear
Arm/Group | Double-blind BTDS 5 | Double-blind BTDS 20 | Double-blind Oxycodone Immediate-Release | Open-label Run-in Period, BTDS 10/20
Serious Adverse Events (participants affected / at risk) | 6/221 | 7/219 | 9/220 | 10/1160
Other Adverse Events (participants affected / at risk) | 54/221 | 118/219 | 93/220 | 389/1160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind BTDS 5 (N=221) | Double-blind BTDS 20 (N=219) | Double-blind Oxycodone Immediate-Release (N=220) | Open-label Run-in Period, BTDS 10/20 (N=1160)
Arrhythmia - DEATH (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Death Systematic and nonsystematic assessments
Brain arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Intractable vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Systematic and nonsystematic assessments
Chest pressure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Worsening chronic cholecycstitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Left lower lobe pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Right heel diabetic foot abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Cocaine toxicity - DEATH (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Death Systematic and nonsystematic assessments
Drowning - DEATH (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Death Systematic and nonsystematic assessments
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Fracture distal right radius (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Herniated disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Clear cell carcinoma left ovary metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Lower extremity lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Lumbar spinal stenosis with diminution of L4-5 (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Nerve entrapment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Depression worsening (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Kidney stones (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Acute bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Acute exacerbation of chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Depressed respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Left pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Diaphoresis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Abdominal aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Hematoma, right thigh (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Acute axonal motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Increased total bilirubin (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Right heel infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind BTDS 5 (N=221) | Double-blind BTDS 20 (N=219) | Double-blind Oxycodone Immediate-Release (N=220) | Open-label Run-in Period, BTDS 10/20 (N=1160)
Nausea (Gastrointestinal disorders) | 18 | 27 | 18 | 174 — Systematic and nonsystematic assessments
Constipation (Gastrointestinal disorders) | 7 | 14 | 14 | 46 — Systematic and nonsystematic assessments
Vomiting NOS (Gastrointestinal disorders) | 5 | 11 | 9 | 60 — Systematic and nonsystematic assessments
Application site erythema (General disorders) | 10 | 22 | 19 | 38 — Systematic and nonsystematic assessments
Application site pruritus (General disorders) | 12 | 29 | 20 | 102 — Systematic and nonsystematic assessments
Application site rash (General disorders) | 17 | 20 | 13 | 38 — Systematic and nonsystematic assessments
Upper respiratory tract infection NOS (Infections and infestations) | 3 | 4 | 10 | 4 — Systematic and nonsystematic assessments
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 10 | 4 | 8 — Systematic and nonsystematic assessments
Headache (Nervous system disorders) | 12 | 25 | 21 | 124 — Systematic and nonsystematic assessments
Somnolence (Nervous system disorders) | 4 | 10 | 11 | 67 — Systematic and nonsystematic assessments
Dizziness (Nervous system disorders) | 5 | 10 | 8 | 62 — Systematic and nonsystematic assessments
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 7 | 13 — Systematic and nonsystematic assessments

LIMITATIONS AND CAVEATS:
BUP3015 was terminated early due to administrative reasons unrelated to efficacy or safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days